CLINICAL TRIAL: NCT06935344
Title: Evaluation of Polygenic Risk Score for Epithelial OVarian cancEr Risk Prediction and Clinical Outcomes in an Italian Population: the PROVE Study
Brief Title: Evaluation of Polygenic Risk Score for Epithelial OVarian cancEr Risk Prediction: the PROVE Study
Acronym: PROVE
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Boccia Stefania, Full Professor of Hygiene and Preventive Medicine, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7225
Record Dates: First submitted 2025-04-09; First posted 2025-04-20 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer
Keywords: polygenic risk score; ovarian cancer; case-control
MeSH Terms: conditions — Ovarian Neoplasms; Genetic Risk Score

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASES: women with ovarian cancer: Patients with histologically proven epithelial ovarian and fallopian tube cancer (referred to as cases), consecutively enrolled in the Ovarian Carcinoma Complex Operative Unit of Policlinico Gemelli.
  Interventions: Genetic: Polygenic Risk Score
- CONTROLS: Healthy women: Women with no previous or concomitant personal history of OC (referred as controls), consecutively enrolled in the Rheumatology Complex Operative Unit of Policlinico Gemelli.
  Interventions: Genetic: Polygenic Risk Score

INTERVENTIONS:
Genetic: Polygenic Risk Score — For the PRS analysis, SNPs for genotyping will be selected based on the latest findings from GWAS on EOC, particularly leveraging the results, as reported by Dareng et al. (doi:10.1038/s41431-021-00987-7). The PRS will be calculated as a weighted sum of risk alleles based on the selected SNPs.

SUMMARY:
The goal of this observational study is to evaluate whether polygenic risk score (PRS) assessment can help predict the onset of epithelial ovarian cancer in women aged over 18, comparing those with a histologically confirmed diagnosis of epithelial ovarian or fallopian tube cancer (cases) to women with no personal history of ovarian cancer (controls). The main questions it aims to answer are:

* Is there an association between PRS and the presence of epithelial ovarian cancer?
* Can PRS improve the prediction of ovarian cancer risk when adjusted for other clinical factors?

Researchers will compare PRS values between cases and controls to see if higher PRS percentiles are associated with an increased risk of ovarian cancer.

Participants will:

* Complete a questionnaire on socio-economic status, lifestyle, and dietary habits.
* Undergo blood sampling, for the analysis of BRCA1-2, PALB2, RAD51C, RAD51D pathogenic variants.
* Undergo PRS analysis.

ELIGIBILITY:
Inclusion Criteria:

* For cases: women with a first-time diagnosis of histologically confirmed epithelial ovarian or fallopian tube cancer.
* For Controls women with no concomitant or past OC diagnosis.

Exclusion Criteria:

* For both cases and controls: the presence of concurrent malignancies other from OC.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer is specific for women
Study Population: Cases and controls enrolment will be conducted in the ovarian cancer and rheumatology outpatient clinics of the Fondazione Policlinico Universitario Agostino Gemelli IRCCS, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Odds of developing EOC by different PRS percentiles | At enrollment
  Correlation between PRS percentiles and EOC risk

SECONDARY OUTCOMES:
Correlation of PRS percentiles and covariates | At enrollment
  Correlation between PRS percentiles and: age, familiarity with OC, stage, histotype, grading (1-2 versus 3), BRCA1-2, PALB2, RAD51C, RAD51D, FANCM status, type of surgery, residual tumor (RT) at histology, type of chemotherapy, maintenance, chemo-resistance, response to treatment, recurrences, progressions, cancer-specific deaths, Disease Free survival (DFS) hazard ratio (HR), Overall Survival (OS) HR.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento Universitario di Scienze della Vita e Sanità Pubblica, Roma, Italia, Italy

IPD SHARING:
Plan to Share IPD: No